CLINICAL TRIAL: NCT03013725
Title: The Hordaland Health Studies (HHS)
Brief Title: The Hordaland Health Study
Acronym: HUSK
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Part of CONOR, and participates in the Norwegian Epidemiologic Osteoporosis Studies (Unknown)
Responsible Party: Principal Investigator, Grethe Seppola Tell, Professor, University of Bergen
Other Study IDs: HUSK9799
Record Dates: First submitted 2016-12-19; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples are stored at two biobanks located in Bergen and Levanger. The blood was divided in full blood, plasma and serum.

GROUPS / COHORTS (2):
- The Homocysteine Study: Conducted in 1992-93, ca. 18000 participated.
  Interventions: Other: No intervention
- The Hordaland Health Study (HUSK): Conducted in 1997-99, ca. 26000 participated.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The Hordaland Health Studies (HHS) were conducted in 1992-93 (The Homocysteine study) and in 1997-99 (HUSK). Both surveys were conducted as a joint project between the University of Bergen, the Norwegian Health Screening Service (SHUS) (now part of the National Institute of Public Health) and the Municipal Health Service in Hordaland.

The main focus of the studies is on chronic diseases including cardiovascular disease, cancer, osteoporosis, anxiety and depression. Some projects focus on psychosocial factors, occupational research, musculoskeletal diseases, urinary incontinence and mapping of drug use. The main purpose of the surveys is to gather information so that disease ultimately can be prevented.

Approximately 36,000 residents of Hordaland county participated in the studies, ca. 18,000 in 1992-93 and ca. 26,000 in 1997-99. About 7,000 of those who participated in the 1992-93 survey also participated in 1997-99.

ELIGIBILITY:
Inclusion Criteria:

* Born in a specific time-period
* From Hordaland County
* Community-dwelling people who were able to come to the study site on their own, and able to fill out questionnaires.

Exclusion Criteria:

* Not born within the specific time-period
* Not from Hordaland County
* Institutionalized People
* People who were not able to fill out questionnaires

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 36,000 residents of Hordaland county participated in the studies (both men and women), ca. 18,000 in 1992-93 and ca. 26,000 in 1997-99. About 7,000 of those who participated in the 1992-93 survey also participated in 1997-99.
Sampling Method: Probability Sample
Enrollment: 36000 (Actual)
Dates: Start 1992-01; Primary Completion 1999-06 (Actual); Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
Total mortality. | Participants are followed from baseline (1992-93 or 1997-99) until death or December 31st, 2015.
  The unique 11-digit personal identification number assigned to all Norwegian residents facilitates linkage between HHS and the Norwegian Population Register, which contains information on vital status (alive, emigrated, or dead). The follow-up period varies from 16 - 23 years, depending on whether first or second measurement is used as baseline.

SECONDARY OUTCOMES:
Mortality or morbidity from chronic diseases (for example cardiovascular disease, cancer). Also, award of disability pension are used as an outcome. | Participants are followed from baseline (1992-93 or 1997-99) until time of diagnosis/death from disease or the last day of follow-up.
  The Cause of Death Registry, Cancer Registry of Norway, CVDNOR and FD-trygd (a national database of Health and social benefits) will be used to get information on outcomes. The last day of follow-up for cardiovascular disease is December 31st, 2014. The last day of follow-up for cancer is December 31st, 2014.
  The last day of follow-up for Cause of Death is December 31st, 2014. The follow-up period for cardiovascular disease varies from 15 - 22 years, depending on whether first or second measurement is used as baseline.
  The follow-up period for cancer varies from 15 - 22 years, depending on whether first or second measurement is used as baseline.

REFERENCES:
- [Derived] Haugsgjerd TR, Egeland GM, Nygard OK, Vinknes KJ, Sulo G, Lysne V, Igland J, Tell GS. Association of dietary vitamin K and risk of coronary heart disease in middle-age adults: the Hordaland Health Study Cohort. BMJ Open. 2020 May 21;10(5):e035953. doi: 10.1136/bmjopen-2019-035953. PMID 32444431
- [Derived] Zuo H, Tell GS, Ueland PM, Nygard O, Vollset SE, Midttun O, Meyer K, Ulvik A. The PAr index, an indicator reflecting altered vitamin B-6 homeostasis, is associated with long-term risk of stroke in the general population: the Hordaland Health Study (HUSK). Am J Clin Nutr. 2018 Jan 1;107(1):105-112. doi: 10.1093/ajcn/nqx012. PMID 29381795